CLINICAL TRIAL: NCT05831449
Title: A Phase 3, Randomized, Double-Blind, Placebo- and Active-Controlled Study to Evaluate the Efficacy and Safety of CPL-01 in the Management of Postoperative Pain After Unilateral Distal First Metatarsal Bunionectomy With Osteotomy
Brief Title: CPL-01 in the Management of Postoperative Pain After Bunionectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cali Pharmaceuticals LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CPL-01-302
Record Dates: First submitted 2023-04-03; First posted 2023-04-26 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Bunion
MeSH Terms: conditions — Bunion | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CPL-01 (Experimental): Local infiltration of study drug
  Interventions: Drug: Local anesthetic injection of CPL-01
- Ropivacaine HCl (Active Comparator): Local infiltration of study drug
  Interventions: Drug: Naropin, 0.5% Injectable Solution
- Placebo (Placebo Comparator): Local infiltration of study drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Local anesthetic injection of CPL-01 — Local anesthetic injection (either IP, positive control [Naropin], or negative control [saline placebo])
  Other Names: CPL-01; Long-acting ropivacaine
  Arms: CPL-01
Drug: Naropin, 0.5% Injectable Solution — Local anesthetic injection (either IP, positive control [Naropin], or negative control [saline placebo])
  Other Names: ropivacaine HCl
  Arms: Ropivacaine HCl
Drug: Placebo — Local anesthetic injection (either IP, positive control [Naropin], or negative control [saline placebo])
  Other Names: Saline placebo
  Arms: Placebo

SUMMARY:
Subjects receive study drug during bunionectomy and are followed for pain and opioid use, with the hypothesis that those who receive CPL-01 will have less pain and less opioid use than either control arm.

DETAILED DESCRIPTION:
After signing informed consent, subjects will be randomly assigned to receive study drug (either Investigational product, positive control, or negative control) during unilateral distal bunionectomy with osteotomy. Subjects will then remain at the hospital for 72-hours where pain and rescue medication usage will be assessed. Follow-up will then occur at 7 and 30 days afterwards.

The hypothesis is that subjects who receive CPL-01 will have less pain and require fewer opioids than subjects in the other two arms.

ELIGIBILITY:
Inclusion Criteria:

* Ability to sign ICF
* Bunion for elective primary unilateral, distal, first metatarsal bunionectomy with osteotomy and internal fixation under regional anesthesia, without collateral procedures or additional surgeries
* BMI ≤ 39 kg/m2
* If biologically female, not pregnant or planning to become pregnant over the study
* If biologically male, either sterile or using acceptable form of birth control
* Be willing and able to complete study procedures

Exclusion Criteria:

* Has previously undergone unilateral simple bunionectomy.
* Has a planned concurrent surgical procedure
* Has a concurrent painful condition that may require analgesic treatment during the study period or may confound postsurgical pain assessments
* Has a history or clinical manifestation of significant medical, neuropsychiatric, or other condition that could preclude or impair study participation or interfere with study assessments.
* Has a history of malignant hyperthermia or glucose-6-phosphate dehydrogenase deficiency.
* Has history or evidence of impaired liver function (e.g., alanine aminotransferase [ALT] > 3 × upper limit of normal [ULN] or total bilirubin > 2 × ULN), active hepatic disease, or cirrhosis.
* Has history or evidence of impaired renal function (e.g., creatinine > 1.5 × ULN).
* Has a history of malignancy in the past year
* Has known or suspected daily use of opioids for 7 or more consecutive days within the previous 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative Pain Score | 72 hours
  Area Under the Curve of the Numeric Rating Scale Score for Pain with Activity. Activity is resting the operative foot with the ball on the floor. Pain Score spans from 0 to 10, where 0 is no pain and 10 is worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Erol Onel, Study Director — Cali Biosciences
Locations (1):
- Todd Bertoch, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No